CLINICAL TRIAL: NCT00005819
Title: A Phase I Trial of Fenretinide in Combination With Paclitaxel and Cisplatin
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Scot C. Remick, MD, : Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU3Y99; U01CA062502 (NIH); P30CA043703 (NIH); CWRU-3Y99 (Other: Case Comprehensive Cancer Center); NCI-T99-0098; CASE-3Y99 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2010-06-11 (Estimated); Status verified 2010-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Cisplatin; Fenretinide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cisplatin — Patients receive cisplatin IV over 30 minutes on day 7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.Cohorts of 3-6 patients receive escalating doses of paclitaxel and cisplatin until the maximum tolerated dose (MTD) is determined.
Drug: fenretinide — Patients receive oral fenretinide twice daily for 7 days. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Other Names: fenretinimide
Drug: paclitaxel — Patients receive paclitaxel IV over 3 hours. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.Cohorts of 3-6 patients receive escalating doses of paclitaxel and cisplatin until the maximum tolerated dose (MTD) is determined.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of combination chemotherapy in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of the combination of fenretinide, paclitaxel, and cisplatin in patients with advanced solid tumors.
* Determine the effect of fenretinide on the pharmacokinetics of paclitaxel and cisplatin.
* Assess the relationship between dose or plasma levels of fenretinide and the safety and antitumor effects, in terms of overall response, response rate, and progression-free survival rate, in these patients.

OUTLINE: This is a dose-escalation study of paclitaxel and cisplatin.

Patients receive oral fenretinide twice daily for 7 days. Patients receive paclitaxel IV over 3 hours and cisplatin IV over 30 minutes on day 7. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of paclitaxel and cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive paclitaxel and cisplatin at the recommended phase II dose.

PROJECTED ACCRUAL: Approximately 15-24 patients will be accrued for this study within 12-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor not amenable to conventional surgery, radiotherapy, or chemotherapy
* No brain metastases or primary brain tumors

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin greater than 9.0 g/dL

Hepatic:

* Bilirubin less than 1.6 mg/dL
* AST and ALT less than 2 times upper limit of normal
* PT and PTT normal OR
* INR less than 1.1

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No extensive signs of macular degeneration, including exudative or atrophic macular lesions reducing corrected vision to less than 20/40

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* Prior platinum-containing agents and taxane exposure allowed with no evidence of neurotoxicity

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered

Surgery:

* Not specified

Other:

* No concurrent vitamin A supplements
* No concurrent supplemental antioxidants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2000-04; Primary Completion 2005-05 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Cohorts of 3-6 patients receive escalating doses of paclitaxel and cisplatin until the maximum tolerated dose (MTD) is determined. | Courses (7 days) repeat every 21 days in the absence of disease progression or unacceptable toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Scot C. Remick, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Locations (1):
- Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States